CLINICAL TRIAL: NCT01903967
Title: Identification of GENEtic Markers of Aggressiveness and Malignancy by Array Comparative Genomic Hybrization Analysis (CGH)
Acronym: PITUIGENE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50834
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Pituitary Tumors
Keywords: Pituitary; CGH array; Tumor
MeSH Terms: conditions — Pituitary Neoplasms; Pituitary Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Pituitary tumour DNA may be extracted from frozen or paraffin-embedded tumours.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- "Control" Group: Patients cured with no evidence of disease up to 5 years will be the controls.
- "Case" Group: Patients, in recurrence or progression before 5 years will be the cases

SUMMARY:
Recent studies estimate that the prevalence of pituitary adenomas is approximately 1/1500 persons. Pituitary tumours are usually considered as benign. However, local invasion is reported in 35-40% of pituitary adenomas; resistance to medical treatment or recurrence leading to multimodal therapy is reported in about 15% of cases. These tumours are considered as aggressive pituitary tumours and present a distinct biological and clinical entity with continued growth despite multimodal therapy, including surgery and radiotherapy (McCormack et al., 2011). Whilst these tumours have malignant potential, the term of pituitary carcinoma is strictly reserved for those rare tumours (0.2%) with demonstrated craniospinal or systemic metastases (Heaney, 2011).

Pituitary aggressive and malignant tumours are very difficult to control and ultimately prove to be lethal. It was suggested that early aggressive treatments (chemotherapy, radiotherapy) may control progression and occurrence of metastases. However, these therapeutic options are associated with important side effects limiting their use and the prediction of pituitary tumor behaviour remains a challenge. At the diagnosis, clinical signs are not specific and the results concerning proliferative factors (Ki-67 and P53), putative oncogenes (PTTG) conflict from one series to another.

In a case-control retrospective study of a cohort of 410 patients (HYPOPRONOS), we validated a prognostic pathological classification based on histological and radiological data (J. Trouillas 2012 in preparation). Tumours were classified into 3 grades: grade 1= non-invasive tumour, grade 2= invasive tumour and grade 3 = aggressive-invasive tumor with the combination of radiological signs of invasion and 2 of 3 signs of increased proliferation (Ki-67 index>3%, number of mitoses>2 per 10 fields at 400X, P53 nuclear detection).

It is now widely accepted that cancer is a clonal disease, which arises from a single normal cell and progresses thanks to the accumulation of DNA alterations (Sanson et al., 2011). To identify the role of these DNA alterations, we conducted array CGH analysis limited to 13 prolactin pituitary tumours, from frozen fragments, and identified allelic loss of chromosome 11 associated with aggressiveness and malignancy (Wierinckx et al., 2011).

To confirm these encouraging results we propose to conduct a study on a large series of tumours, fixed and embed, and to be correlated the results to clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Only patient with complete clinical, radiological and hormonal data available during yearly follow-up will be included.
* Preoperative MRI will be used to classify the tumour as invasive, and postoperative MRI will be collected to confirm recurrence or progression of the tumour.
* Presence of tumour fragments fixed in Holland-Bouin's fluid or Neutral Buffered Formalin fixative available for aCGH analysis.

Exclusion Criteria:

* Patient who underwent systematic post-operative radiotherapy.
* Patient presenting Multiple Endocrine Neoplasia type 1 (MEN1) or aryl hydrocarbon receptor interacting protein (AIP) mutation since mechanism of tumorigenesis are different to sporadic pituitary tumours.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting a pituitary tumour, including PRL, GH, ACTH and LH/FSH, operated on by transsphenoidal route between 1990 and 2008 with at least 5 years of follow-up
Sampling Method: Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2013-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
DNA alterations associated with the prognosis of pituitary tumours. | At least 5 years of follow-up
  To identify and quantify the genomic DNA alterations associated with the prognosis of pituitary tumours.

CONTACTS AND LOCATIONS:
Overall Officials: Gérald RAVEROT, PhD - MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Groupement Hospitalier Est, Lyon, France

REFERENCES:
- [Derived] Lasolle H, Raverot G. Letter to the Editor From Helene Lasolle and Gerald Raverot: "USP8 and TP53 Drivers Are Associated With CNV in a Corticotroph Adenoma Cohort Enriched for Aggressive Tumors". J Clin Endocrinol Metab. 2021 Jul 13;106(8):e3285-e3286. doi: 10.1210/clinem/dgab217. No abstract available. PMID 33822961
- [Derived] Lasolle H, Alix E, Bonnefille C, Elsensohn MH, Michel J, Sanlaville D, Roy P, Raverot G, Bardel C. Centralization errors in comparative genomic hybridization array analysis of pituitary tumor samples. Genes Chromosomes Cancer. 2018 Jun;57(6):320-328. doi: 10.1002/gcc.22534. Epub 2018 Mar 9. PMID 29460398
- See also: Related Info — http://federation-endocrino-poleest.univ-lyon1.fr